CLINICAL TRIAL: NCT02146443
Title: Validation and Test-retest Study of the Star-shaped Manual Dexterity Test.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Niels Kildebro, BSc.med., Scholar student, Herlev Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: STAR-222
Record Dates: First submitted 2014-05-21; First posted 2014-05-23 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Manual Dexterity
Keywords: Manual dexterity; hand to eye coordination; stress; fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Baseline (Active Comparator): Completion of the star shaped manual dexterity test, five rounds clockwise and five rounds counter clockwise without any intervention. Time and number of errors are recorded. Measurement of static arm strength with the stretched arm test. test subject is asked to hold a 2.5 kg weight in stretched arm for as long as possible. Maximum endurance time is recorded.
  Interventions: Other: Stretched arm test; Device: Star shaped manual dexterity test
- Fatigue (Active Comparator): Prior to completion of the star shaped manual dexterity test, the test subject is asked to stand up still and hold a 2.5-kg weight with the dominant arm fully extended as long as possible without moving. Maximum endurance time is recorded. After this, the test subject completes the the star shaped manual dexterity test and time and number of errors are recorded.
  Interventions: Other: Stretched arm test; Device: Star shaped manual dexterity test
- Stress (Active Comparator): During completion of the star shaped manual dexterity test, the test subject is asked to identify cards from a regular deck of playing card by naming the suit and rank of the card. They will be asked to identify one random card during each of the 10 rounds in the completion of the test. Completion time and number of errors are recorded.
  Interventions: Other: Stress; Device: Star shaped manual dexterity test
- Fatigue and Stress (Active Comparator): The test subject will be fatigued prior to the test (as detailed in the fatigue arm), and asked to identify cards during completion of the star shaped manual dexterity test (as detailed in the stress arm). Completion time and number of errors are recorded.
  Interventions: Other: Stretched arm test; Other: Stress; Device: Star shaped manual dexterity test

INTERVENTIONS:
Other: Stretched arm test — Measurement of static arm strength. Test subject is asked to hold a 2.5 kg weight in their dominant arm fully extended at 90-degree flexion and 15-degree abduction as long as possible without moving.
  Arms: Baseline; Fatigue; Fatigue and Stress
Other: Stress — During completion of the star shaped manual dexterity test, the test subject is asked to identify cards from a regular deck of playing card by naming the suit and rank of the card. They will be asked to identify one random card during each of the 10 rounds in the completion of the test
  Arms: Fatigue and Stress; Stress
Device: Star shaped manual dexterity test — On a piece of wood, a piece of metal (dimensions 22 cm x 22 cm) is mounted. In the center of the metal plate, is a star shaped track. The star has 6 points and the track is 9 mm wide. It measures 15,3 cm from the tips of opposing arms of the star. With a surgical scissor in his dominant hand, the test subject is instructed to follow the star shaped track ten times, five times clockwise and five times counter clockwise. Contact with the border of the track is counted as an error. A computer software program automatically registers completion time and number of errors. The test is conducted in an undisturbed environment.

SUMMARY:
The purpose of this study is to measure test-retest reliability and validate the star shaped test of manual dexterity. The purpose of this is to see if there is any significant learning effect, and if the test can discriminate between individuals who are at their normal skill level, and when they are stressed and/or fatigued. The test is designed to test hand to eye coordination and precision control. This is done by following a star shaped track with a pair of a surgical scissors. this is done 10 times, 5 times clockwise and 5 times counter clockwise. Each time the scissors come into contact with the border of the track, an error is counted. Overall completion time is recorded. As a randomized crossover study, we will have 20 test subjects complete the test 4 times. Each test will be conducted with a pause of two breaks between the tests. Before each test, the test subjects are randomized to: no intervention, physical fatigue prior to testing, distractions during the test or both physical fatigue prior to testing and distractions during the test. All participants will complete a test with all four interventions. Furthermore, a test-retest trial will be conducted on 4 test-subjects. Each subject will complete the test two times with no interventions, with two days apart.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 55 years

Exclusion Criteria:

* Diagnosed heart disease
* Diagnosed endocrinological disease
* Diagnosed Neurological or autoimmune disease
* Diagnosed Sleep disorder
* Diagnosed orthopedic diseases or former orthopedic surgery (e.g. arthrosis, rotator cuff syndrome)

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2014-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Completion time of the star shaped manual dexterity test. | up to day 10
  The time in seconds it takes to complete 10 rounds of the star shaped manual dexterity test. First 5 rounds clockwise and then 5 rounds counter clockwise. The test will be performed on day 1, 4, 7 and 10 of the study.

SECONDARY OUTCOMES:
Number of errors during the completion of the star shaped manual dexterity test. | Test completion period at day 1, 4, 7 and 10
  An error is counted each time the test subject touches the borders of the star shaped track of the manual dexterity test with the surgical scissor.

CONTACTS AND LOCATIONS:
Overall Officials: Niels Kildebro, BSc.med., Principal Investigator — Herlev Hospital, Copenhagen University
Locations (1):
- Herlev Hospital, Herlev, Herlev, Denmark